CLINICAL TRIAL: NCT03820310
Title: Clinical Trial of Autologous Tcm Cellular Immunotherapy Combined With Traditional Therapy in Intrahepatic Cholangiocarcinoma Patients After Radical Resection
Brief Title: Clinical Trial of Autologous Tcm Immunotherapy in ICC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newish Technology (Beijing) Co., Ltd. (Industry)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-IT-004
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cholangiocarcinoma
Keywords: malignancy; intrahepatic cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): traditional therapy plus autologous Tcm cellular immunotherapy.
  Interventions: Biological: autologous Tcm cellular immunotherapy
- control group (No Intervention): traditional therapy alone, such as radiotherapy or chemotherapy.

INTERVENTIONS:
Biological: autologous Tcm cellular immunotherapy — autologous cellular immunotherapy plus traditional therapy. • cells will be infused in 3-5×109 cells/100 ml 1 month after radical resection, then cells will be infused as the same dose followed by a 1 month rest period, Each subject in experimental group will receive a total of 5 cell infusions.
  Arms: Experimental group

SUMMARY:
The prime purpose of this trial is to evaluate the Progression Free survival and two-year survival of combining autologous Tcm cellular immunotherapy and traditional therapy in intrahepatic cholangiocarcinoma (ICC) patients after radical resection. A secondary objective of the trial is to assess the long-term survival and safety of Tcm cellular immunotherapy and traditional therapy in ICC patients after radical resection. Patients will be randomized 1:1 either to the experimental group to receive autologous Tcm cellular immunotherapy and chemotherapy or to the control group (traditional therapy).

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (ICC) accounts for 2%~3% of gastrointestinal tumors, and the incidence has been on the rise globally. The pathogenesis of ICC remains unclearly. Compared with palliative resection, the postoperative survival rate of patients undergoing radical resection is significantly improved. However, most patients after radical resection will recurrence or metastasis, and the five-year overall survival rate is about 10-40%.

Autologous cellular immunotherapy is to collect patient's own immune cells and infuse into the patient's body after culture in vitro that can activate the anti-tumor immune response and then achieve the purpose of cancer treatment. Central memory T cells (Tcm) is the most effective anti-tumor immune cell with long-term in vivo survival and self-renewal capacity. Combination of autologous cellular immunotherapy with traditional therapies, such as radiotherapy or chemotherapy, can effectively prolong the survival period of patients, and improve the quality of life for patients.

This study will recruit subjects with pathologically confirmed intrahepatic cholangiocarcinoma after radical resection. Patients must have adequate hematologic and end organ function, performance status and no contraindications to receive autologous cellular immunotherapy.

The observation period of patients is 24 months. The prime purpose of this trial is to evaluate the Progression Free Survival (PFS) and two-year survival of combining autologous Tcm cellular immunotherapy and traditional therapy in intrahepatic cholangiocarcinoma (ICC) patients after radical resection. A secondary objective of the trial is to assess the long-term survival and safety of Tcm cellular immunotherapy and traditional therapy in ICC patients after radical resection.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial
2. Subjects treated with radical resection completely, and pathologically confirmed intrahepatic cholangiocarcinoma
3. Subjects with image examination confirmed complete response (CR) postoperatively
4. Age between 18 and 70 years old
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Normal hematopoietic function:

   White Blood Cell (WBC) ≥ 4×10^9 /L Neutrophil ≥ 2×10^9 /L Hemoglobin ≥ 90 g /L Platelets ≥ 100×10^9 /L
7. Lymphocyte ≥ 0.7×10^9 /L
8. Adequate Liver and kidney function Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 the upper limit of normal (ULN) for the institution Total bilirubin (TBIL) ≤ 1.5 the upper limit of ULN Serum creatinine (CREA) ≤ 1.5 the upper limit of ULN Creatinine clearance ≥ 70 ml/min
9. Subjects without significant cardiovascular and lung disease

Exclusion Criteria:

1. Subjects with recurrent intrahepatic cholangiocarcinoma
2. Subjects who are using immunosuppressive agents or long-term immunosuppressive agents after organ transplantation.
3. Subjects with severe abnormality of coagulation;
4. History or any evidence of hemorrhage.
5. Subjects with bone marrow transplant or severe leukopenia
6. Subjects with severe heart, liver or kidney diseases.
7. Subjects with severe infection or high fever.
8. Subjects with severe autoimmune diseases.
9. Subjects infected with HIV
10. Subjects combined with other malignancies
11. Subjects with T-cell lymphma or tumor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 24 months
  The Progression Free Survival of combining autologous Tcm cellular immunotherapy and traditional therapy in ICC subjects after radical resection.
Two-year survival | 24 months
  Two-year survival of combining autologous Tcm cellular immunotherapy and traditional therapy in ICC subjects after radical resection.

SECONDARY OUTCOMES:
The long-term survival of ICC subjects | 24 months
  The long-term survival of ICC subjects treated with Tcm cellular immunotherapy and traditional therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Shunda Du, M.D, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No